CLINICAL TRIAL: NCT04451512
Title: A Prospective Observational Study of Cold and Hot Snare Resection for Colorectal Polyps Sized 10-19mm.
Brief Title: Comparison of Cold and Hot Snare Resection for Colorectal Polyps Sized 10-19mm.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 20200615
Record Dates: First submitted 2020-06-17; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Colonic Polyps/Colonoscopy/Colorectal Neoplasms
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colorectal polyps after resection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSP
- HSP

SUMMARY:
Patients who met the criteria for removal of 10-19mm colorectal polyps using cold snare or hot snare were included in the study, signed by endoscopic treatment written informed consent for surgery, patients with detailed tracking and record the basic information and information related to the operation, postoperative lack of region and edge endoscopic observation carefully no residue, additional excision may be took if necessary，after resection specimen inspection, and in 6 months review colonoscopy, assess whether there is residual or recurrence of polyps.Main outcome: technical success rate (no other auxiliary resection), complete resection rate, secondary outcome: intraoperative and postoperative complications, polypectomy time and related costs, influential factors of incomplete resection.Research significance: The effectiveness, safety and cost-effectiveness of cold and hot snare resection of 10-19mm colorectal polyps were compared, and the influencing factors of incomplete polyps resection were analyzed, so as to provide evidence for the decision on the best method of medium-size polyps resection.

ELIGIBILITY:
Inclusion Criteria:

1. colorectal polyps sized 10≤ diameter ≤19 mm;
2. Boston bowel prepare score: 5-9;
3. The patients all signed the informed consent of endoscopic treatment.

Exclusion Criteria:

1. Complicated with inflammatory bowel disease, P-J syndrome or familial polyposis;
2. Complicated with malignant tumors;
3. polyp size is uncertain;
4. Currently taking aspirin, warfarin or other anticoagulants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the criteria for removal of 10-19mm colorectal polyps using cold snare or hot snare were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | 2020.07.31
  (without other auxiliary resection)
Complete resection rate | 2021.01.31

SECONDARY OUTCOMES:
Intraoperative and postoperative complications | 2021.01.31
Polypectomy time | 2021.01.31
related costs of treatment | 2021.01.31

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided